CLINICAL TRIAL: NCT00900497
Title: A Phase I/II Study For the Use of White Blood Cells From Healthy Donor-participants To Treat Subjects With Solid Cancers
Brief Title: A Study Using White Blood Cells From Healthy Donors To Treat Solid Cancers
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dipnarine Maharaj (Other)
Responsible Party: Sponsor-Investigator, Dipnarine Maharaj, Medical Director, South Florida Bone Marrow/Stem Cell Transplant Institute
Organization: South Florida Bone Marrow/Stem Cell Transplant Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08001-BMSCTI
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumors
Keywords: granulocytes; Graft-vs-Host-Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Leukocyte Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- White Blood Cells/Granulocytes (Experimental): Fresh, non-irradiated granulocytes from ABO-Rh compatible, HLA-mismatched donors
  Interventions: Biological: White Blood Cells/Granulocytes

INTERVENTIONS:
Biological: White Blood Cells/Granulocytes — Granulocytes collected by apheresis, cross-matched for ABO-Rh and common antibodies, HLA-mismatched to avoid engraftment

SUMMARY:
Background & Rationale:

About 75% of US population living today will not die of cancer. There has been a recent report of a colony of cancer-resistant mice developed from a single male mouse that unexpectedly survived challenges of lethal cancer cell injections. In these so-called spontaneous regression/complete resistant (SR/CR) mice, cancer cells are killed by rapid infiltration of leukocytes, mainly of innate immunity. This highly effective natural cancer immunity is inherited and mediated entirely by white blood cells. Moreover, this cancer resistance can be transferred to wild type mice through the transfer of various immune cell types including granulocytes. The infusion of white blood cells, particularly cells of innate immunity, is a viable anticancer therapy in humans as well. This proposed trial will test whether white blood cell infusions from healthy unrelated donors can be used to treat cancer. The trial is designed to determine whether responses can be seen in cancer patients after infusion of HLA-mismatched white cells from healthy donors. It is important that the donors and recipients be unrelated and HLA-mismatched to avoid the possibility of transfusion-related Graft vs. Host Disease. The white blood cells from the healthy donors are being collected via apheresis following granulocyte mobilization with dexamethasone and filgrastim. The investigators will refer to the white blood cells as 'granulocytes' because 75-90% of the white blood cells collected through the apheresis will consist of granulocytes. The dose of at least 2x10 to the11th will be given from 4-5 donors at a rate of no more than one donor per day for each recipient. There will only be one infusion per day and no more than 5 infusions per week. Thus, a typical treatment in the study would span 1-2 weeks. After each infusion, the patients will be monitored carefully for possible adverse events. If adverse events occur at any time point during or after individual infusion, the treatment can be stopped until the adverse events can be managed. The daily dose of each infusion is a frequently used level that has a long safety record. The trial will observe the subject's cancer for 3 months after the granulocyte infusions are completed. Response at 90 days will be based on comparison of tumor measurements at baseline. The trial has 3 major endpoints: dose response and tolerance, safety, and efficacy.

DETAILED DESCRIPTION:
Up to 29 Subjects with metastatic, non-hematological cancer can be entered. Potentially hundreds of healthy Donor-participants will be recruited. A Donor Registry will be built to store ABO/Rh-specific donors; these donors will be tested for HLA-specific genotyping as well as fully tested for infectious diseases.

Each patient will be receiving granulocytes from approximately 4 to 6 donors. Each donor will be HLA-mismatched to avoid engraftment of the granulocytes and any transfusion-related GVHD. These infusions will take place over a 1 to 2 week period, the timing of which will be dependent on both the subject's tolerance and the availability of the donors.

Subject Response Assessment:

For all patients not demonstrating disease progression, response status will be evaluated between Days +90 to +100 after the last infusion. Day+1 is the first day of white cell infusion. All measurable lesions (lesions that can be accurately measured in at least one dimension [longest diameter to be recorded] as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan) up to a maximum of 10 lesions representative of all involved organs should be identified as target lesions and will be recorded and measured at baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repetitive measurements (either by imaging techniques or clinically). A sum of the longest diameter (LD) for all target lesions will be calculated and reported as the baseline sum LD. The baseline sum LD will be used as reference to further characterize the objective tumor response of the measurable dimension of the disease. The criteria for response, progression, and relapse are as follows.

* Complete Response: Disappearance of all target lesions.
* Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
* Progression (PD): At least a 20% increase in the sum of the LD of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
* Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD since the treatment started. Patients having a documented response with no reconfirmation of the response will be listed with stable disease.

ELIGIBILITY:
Inclusion Criteria for Subjects:

* Must have signed Subject Informed Consent form
* Documentation of Disease: All patients must have histologically or cytologically confirmed non-hematological malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Measurable Disease: Lesions that can be accurately measured in at least one dimension (longest diameter recorded) as ³20 mm with conventional technique or as ³10 mm with spiral CT scan.
* Life expectancy of at least 4 months as judged by the PI at the time of consent
* Performance status of ≤2 on the ECOG scale (see Appendix I).
* ≥ 4 weeks since prior medical therapy, radiation therapy, and surgery
* Adequate organ function, such as absolute neutrophils ≥1,500/µl, platelet transfusion independent,
* platelet count ≥100,000/µl, serum bilirubin ≤2 mg/dl, AST/ALT less than 3x upper limit of normal and serum creatinine ≤2 mg/dl.

Exclusion criteria:

* Uncontrolled diabetes mellitus, significant cardiac disease, e.g. recent myocardial infarction ≥ within 30 days, or active serious infection.
* HIV infection and no recent use (within 30 days) of immunosuppressive agents other than steroids.
* Pregnant or nursing women.
* Men or Women of reproductive age who are not using an effective means of birth control.
* Women of childbearing potential who have a positive serum pregnancy test prior to treatment.
* HLA Class I & II antibodies.
* Neutrophil antibody test.
* Prior history of stem cell transplantation.
* Evidence of brain tumors or metastases.
* Prior history of fludarabine therapy.

Inclusion Criteria for Granulocyte Donors:

* Must have signed Donor-participant Informed Consent Form
* Must be a healthy, eligible blood donor who has completed Full-Length Universal Donor History Questionnaire version 1.2
* Must be able to donate granulocytes and be willing to undergo granulocyte apheresis
* Must have an HLA profile (A, B, DR) with results that ensure donated granulocytes will be mismatched with the recipient
* Must have CMV negative or positive sero-testing completed; only seronegative donors are accepted for a seronegative recipient
* Must have compatible ABO and RH typing with the subject
* Must be negative for HLA Class I & II antibodies

Exclusion criteria:

* Positive Neutrophil antibody test
* Positive infectious disease workup within 30 days of apheresis / donation.
* Positive known cardiac illness that could cause a potential risk associated with leukapheresis.
* Genetic relationship to the recipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2009-04; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The trial will observe the subject's cancer status for 3 months after the granulocyte infusions are completed. Response at 90 days will be based on comparison of tumor measurements at baseline. | 90 to 100 days post treatment

SECONDARY OUTCOMES:
The trial will evaluate the safety and dose tolerance of the transfusion of non-irradiated granulocytes (approximately 4 to 6 donors to reach a level of 2 x 10 to the 11th cells) from HLA-mismatched donors | 1 to 2 weeks treatment and 30 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dipnarine Maharaj, MD, Principal Investigator — Medical Director, South Florida Bone Marrow / Stem Cell Transplant Institute
Locations (1):
- South Florida Bone Marrow / Stem Cell Transplant Institute, Boynton Beach, Florida, United States